CLINICAL TRIAL: NCT06957132
Title: Analysis of Risk Factors for Hearing Loss in Survivors of Cancer Occurred During Childhood, Adolescence or Young Adulthood
Acronym: RISP-OTOTOX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-A02705-42; 2024/3979 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2025-04-17; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Ototoxicity, Drug-Induced; Ototoxicity, Radiation-Induced; Pediatric Cancer
MeSH Terms: conditions — Ototoxicity; Neoplasms | interventions — Audiometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Audiologic examination (Other): Add an audiogram in the patient consultation
  Interventions: Device: Audiogram

INTERVENTIONS:
Device: Audiogram — Either the patient can be proposed to perform the audiogram during their long-term consultation, or they will be contacted by the physician to come especially for the project and realize the audiogram.
  iAudiogram is an Artificial Intelligence (AI) - automated audiometry platform (https://iaudiogram.com/), certified CE (European conformity).
  This examination will be performed once within the study.
  Other Names: iAudiogram medical device

SUMMARY:
This study is aimed at people treated for cancer before the age of 25, who have been followed for at least 5 years, and who are now aged between 18 and 50. It is a prospective, multicenter, non-randomized study.

The main aim of the project is to identify hearing impaired patients using the iAudiogram medical device, and to analyze the risk factors associated with the risk of hearing impairment.

Around 500 patients will take part in this study in France. Participation in this research project will consist in carrying out a hearing test (audiogram with tonal audiometry) with the iAudigram medical device (at Gustave Roussy, Curie or Necker Hospital) and completing self-questionnaires focusing on ototoxicity and its consequences.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 50 years at audiological investigations
* Treated for brain tumor, solid cancer, lymphoma or leukemia in childhood, adolescence or at a young adult age (<25years)
* With at least 5 years of cancer-free follow-up after childhood cancer
* Patients included in the FCCSS ( https://fccss.fr ) deep cohort of 7670 5-year childhood cancer survivors treated before 2001, or patients who have planned visit in long-term follow-up clinics of Curie Institute and Gustave Roussy, whatever the diagnostic period
* Pregnant or breast-feeding women can be included as no risk is identified
* With Social security coverage
* Signed written informed consent obtained

NB: Patients included in another research project are not excluded from this one

NB: patients wearing a Lyric hearing prosthesis or any other permanent hearing prosthesis or cochlear implant can be included in the study but will not perform audiological examinations because the audiogram can't be easily performed without hearing prosthesis. Nevertheless, these patients could participate to the study with self-administered questionnaires and could be included as cases (i.e. patients with hearing deficiency) in analyses.

Exclusion Criteria:

* Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent
* Patient with unavailable data concerning treatment modalities including cumulative doses of chemotherapy agents or radiation fields and dose

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
measurement of hearing loss by frequency and/or sound level | Baseline
  The patients explored with the automated tonal audiometry (iAudiogram medical device) with one of the following results as well as patients wearing a Lyric hearing prosthesis or any other permanent hearing prosthesis or cochlear implant will be considered as as having an audiological impairment:
  * Average hearing loss at 500Hz 1kHz 2kHz 4kHz 8kHz, ≥ 30dB
  * Hearing loss at least on 2 adjacent frequencies (among 500Hz 1kHz 2kHz 4kHz 8kHz) ≥ 30dB
  * Hearing loss at 8kHz ≥ 40dB (Brock1, according to Brock Grading system)
  * Asymmetrical hearing: interaural gap of ≥ 15 dB on two adjacent frequencies or interaural gap of ≥ 25 dB on one frequency
  * Abnormal result on high-frequency audiometry: hearing loss at least on 2 points on frequencies 11.2-16 kHz, ≥ 30 dB

CONTACTS AND LOCATIONS:
Overall Officials: Brice Fresneau, MD, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (3):
- France (3):
  - Hôpital Necker, Paris
  - Institut Curie, Paris
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No